CLINICAL TRIAL: NCT04165265
Title: Reduction in Length of Hospitalization in Patients With Acute Severe Ulcerative Colitis Treated With Rescue Therapy With Infliximab by the Use of Web-app Constant-Care. One Year Follow-up, Inclusive Colectomy Rate.
Brief Title: The Use of Web-app Constant-Care in Patients With Acute Severe Ulcerative Colitis Treated With Rescue Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nordsjaellands Hospital (Other)
Collaborators: Calpro AS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-19047104
Record Dates: First submitted 2019-11-08; First posted 2019-11-15 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-11

CONDITIONS: Ulcerative Colitis; Telemedicine
Keywords: Hospitalization; Reduction in stay; Ulcerative Colitis; Inflammatory Bowel Disease; eHealth; Colectomy; Rescue therapy; Infliximab
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Intervention Model Description: Case-control trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Responders and Partial/non-responders (Experimental): The definition of responders to glucocorticoids is: "Bowel movements ≤ 3/day without blood and normalization of CRP". In the study, this is supported by CC.
  The definition of non-responders is: "Bowel movements > 8/day or 3-8/day and CRP > 45 mg/l." The decision if the patient is a non-responder is supported by CC.
  Questionnaires in CC and FC analysis with CalproSmart are performed every day until discharge or when classified as "green" in CC. After discharge questionnaires in CC and FC analysis are performed once every week in the following 7 weeks and a final registration at week 52. In case of disease relapse between week 7 and 52 registration in CC and FC analysis are performed on demand. Fecal samples for future use (biobank) and FC Elisa as well as blood samples are done before administration of IFX (week 2 and 6). At follow-up (week 52) it is considered whether the patient underwent colectomy or not.
  Interventions: Device: Constant-Care

INTERVENTIONS:
Device: Constant-Care — Constant-Care (CC) (https://ibd.constant-care.com) is a web-application and contains an education and a disease monitoring package. An algorithm is established in the disease monitoring package, which consist of two variables; fecal calprotectin (FC) and a disease activity questionnaire (validated), Simple Clinical Colitis Activity index (SCCAI) for UC. The FC is obtained through CalproSmart app (it only takes 18 min) and the questionnaire is filled out in CC. Afterwards, the data are analyzed by CC and presented in a Total Inflammatory Burden Score (TIBS) as well as a visual "traffic light" of disease for the patients

SUMMARY:
The primary aim is to evaluate if introduction of eHealth in its form of the web application Constant-Care (https://ibd.constant-care.com) could reduce the length of hospitalization in patients with acute severe Ulcerative Colitis treated with infliximab. This is relative to historical controls extracted from medical records.

Patients will self-measure on the web-application while hospitalized as well as after discharge. At the web-application different questionnaires are filled out and a fecal calprotectin (FC) analysis is performed on a smartphone. The final follow up is one year after admission.

DETAILED DESCRIPTION:
Consecutive inclusion of patients hospitalized at North Zealand University Hospital (NOH) in Denmark between December 2019 and June 2020 with the diagnosis acute severe Ulcerative Colitis (UC) (expected 14-28 patients). The included patients will be matched with historical controls 1:3 (matched on age and sex). Controls will be extracted from medical records (2015-2019). Only historical controls who meet the inclusion criteria as well as receive Infliximab rescue therapy, when admitted to hospital due to the diagnosis acute severe UC, are included. This means that patients, who are responders to high dose glucocorticoids are excluded as historical controls.

At Day 0 all the included UC patients will receive an introduction and their own personal login to the Constant-Care (CC) web-application (Two Factor Authentication) as well as receive standard treatment with IV glucocorticoids. When the patients have received an introduction to CC, they will register their disease activity; Simple Clinical Colitis Activity index (SCCAI). This tool captures the patient's illness experience (Patient-Reported Outcomes, PROs). Furthermore, the patients are introduced and assisted with Fecal Calprotectin (FC) testing kit (CalproSmart). For this analysis, patients will receive a personal login to CalproSmart.

Beside the CC monitoring initiated at Day 0, the patient will be followed through standard monitoring (DSGH guidelines) such as vital parameters daily (minimum three times a day), conventional FC Elisa (send to Hvidovre), blood samples and the frequency of bowel movements. In addition, fecal samples will be collected from all patients to microbiome analysis for future use (I Suite nr: 03719, ID no: NOH-2015-017). A separate written informed consent is collected when patient want to participate in future research with microbiome analysis. Furthermore, the patients' medical history, disease course and Montreal classification will be examined. At follow-up (week 52) it is considered if the patient had a colectomy.

While hospitalized patients register in CC everyday as well as perform the FC test with CalproSmart. This is continued until discharge or whenever the patient is categorized as "green". A patient is classified as "green" when either SCCAI or FC are in the green zone (cut-off values: SCCAI; ≤ 2 (green), > 2 - 5 (yellow) and > 5 (red), FC; ≤ 200 mg/kg (green), 201-600 mg/kg (yellow), > 600 (red)).

On or around Day 3 it is considered if patient is a responder to the initial treatment with glucocorticoids. In case only partial or no response is observed the patient is considered rescue therapy (Infliximab, IFX) if no contraindications are present. This divides the patients in two arms; responders and partial/non-responders.

Both groups will continue daily registration in CC and perform FC test while admitted to hospital or until classified as "green". After discharge the responder group will register in CC and perform FC on demand in case of relapse in disease. At follow up (week 52) responders will register in CC and perform the FC test.

Partial/non-responders will, after discharge, register in CC and perform FC test once every week in the following 7 weeks. Afterwards registration is done on demand in case of relapse in disease. A final registration in CC and FC test is done at follow up.

In CC, patients will register: SCCAI, S-IBDQ, WEB-DI and FC via CalproSmart.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the diagnosis acute severe UC/IBDU, ECCO guidelines; Bloody diarrhea ≥ 6/day plus minimum one of following: Pulse > 90/min, Temperature > 37.8 °C, Hemoglobin < 105 g/l, ESR > 30 mm/h, CRP > 30
* Hospitalized at NOH, Hillerød
* UC patients receiving IV glucocorticoids
* UC patients who can read, speak and understand Danish
* Have a smartphone
* UC patients who can manage going on Internet
* Above 18 years of age

Exclusion Criteria:

* Any present enteric infection
* Receiving per oral glucocorticoids
* Contraindications for IFX therapy, including;

  1. Former inadequate response to IFX
  2. Disease relapse in spite of current treatment with IFX
  3. Intolerance or unacceptable side-effects to IFX
  4. Active or latent TB
  5. Cardiac failure (NYHA III or IV)
  6. Demyelinating disorders
* Former gastrointestinal surgery
* UC patients with any severe mental disturbance and/or alcohol/other drug abuse
* UC patients with language barrier
* Below 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2019-12-03 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in length of hospitalization due to the use of Constant-Care | One year after inclusion
  The primary aim is to evaluate if introduction of eHealth in its form of the web application Constant-Care could change the length of hospitalization in patients with acute severe Ulcerative Colitis treated with infliximab. This is relative to historical controls extracted from medical records.

SECONDARY OUTCOMES:
Quality of Life (S-IBDQ) | One year after inclusion
  S-IBDQ is a clinical tool, which measure the subjective health related quality of life (HRQoL) in patients with an IBD diagnosis. The questionnaire compromises 10 questions derived from the full version IBDQ. Questions cover patients physical health, psychological health, social relationships and environment. The total score ranges from 10 to 70, where 70 indicates best health (classified as "green" in CC when S-IBDQ > 50). Evidence has shown that the tool is able to discriminate between patients with active and inactive disease. Furthermore, evidence indicates that S-IBDQ correlates with other clinical tools such as the SCCAI.
  Interesting questions concerning the S-IBDQ are: How will the S-IBDQ change over time (responder and non-responder)? What are the differences between responders and non-responders? What is the impact of S-IBDQ in relation to clinical decision-making?
Disability index (WEB-DI), The IBD Disk | One year after inclusion
  The IBD Disk was developed from selected elements from the IBD disability index (IBD-DI), which are most likely to be important in assessing a patient's disease burden and at the same time had relevance to both the patient and physician. The IBD-DI consists of 28 questions and is a physician- administrated tool, which evaluates the IBD patients' functional status. The IBD Disk consists of 10 elements, which are ranked from 0 to 10; Abdominal pain, regulating defecation, interpersonal interactions, education/work, sleep, energy, emotions, body image, sexual functions and joint pain. The result is visually illustrated in a disc.
  Interesting questions concerning the WEB-DI are: How will the WEB-DI change over time (responder and non-responder)? What are the differences between responders and non-responders? What is the impact of WEB-DI in relation to clinical decision-making?
Fecal calprotectin level | One year after inclusion
  FC release is related to cell stress/damage and is a very sensitive marker for inflammation in the gastrointestinal tract. It is available as a non-invasive tool for monitoring and adjustment of treatment in UC as it relates to relapse in the disease. Furthermore, there is a high correlation between FC level measured in stool and the histological and endoscopic findings. In the study FC would be analyzed with conventional FC Elisa and by the use of Calpro Smart
  Interesting questions concerning the fecal calprotectin level are: How will the calprotectin level change over time (responder and non-responder)? What are the differences between responders and non-responders? What is the lead time between fecal calprotectin determination via CalproSmart and conventional Elisa? What is the impact of the immediate calprotectin analysis via CalproSmart to clinical decision-making?
Time to clinical decision-making (days) | One year after inclusion
  The conventional treatment of patients with acute severe UC is IV glucocorticoids. No response to glucocorticoids is associated with colectomy in 85% of cases during the actual admission if rescue therapy is not initiated. Infliximab, which is one of the therapeutic alternatives, has been found safe and effective as rescue therapy (reduction in colectomy rate) in patients with acute moderate to severe UC. The response to the treatment with glucocorticoids is evaluated at Day 3-5. If no or only partial response is observed, it is considered if the patient is a candidate for the rescue therapy with IFX between Day 3 and 5. However, Day 3-5 is rarely being withhold in everyday life in hospital.
  Interesting questions concerning the time to clinical decision-making: Will time to clinical decision-making change relative to historical controls? This would be an estimate relative to the length of hospitalization. What are factors that determine whether to start infliximab or not?
Colectomy rate (at week 52) | One year after inclusion
  Will the colectomy rate change (decrease/increase/unaffected) compared with the historical controls?
Disease course types | One year after inclusion
  The disease course of UC patients is varying. Overall, they are considered in four subgroups characterized based on relations between periods of active disease and remission. The groups are as follows:
  1. High disease activity in the beginning, followed by decreasing disease activity
  2. Low disease activity in the beginning, followed by increasing disease activity
  3. Chronic disease course with constant disease activity
  4. Chronic disease course with fluctuations in disease activity
  Interesting questions concerning disease course types: Are the patients disease course changed over time? Will there be any differences between responders and non-responders? Does the initial disease course have an impact on the outcome of the admission?

CONTACTS AND LOCATIONS:
Overall Officials: Pia Munkholm, Professor, Study Director — North Zealands University Hospital
Locations (1):
- North Zealand University Hospital, Frederikssund, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elkjaer M, Shuhaibar M, Burisch J, Bailey Y, Scherfig H, Laugesen B, Avnstrom S, Langholz E, O'Morain C, Lynge E, Munkholm P. E-health empowers patients with ulcerative colitis: a randomised controlled trial of the web-guided 'Constant-care' approach. Gut. 2010 Dec;59(12):1652-61. doi: 10.1136/gut.2010.220160. PMID 21071584
- [Background] Pedersen N, Thielsen P, Martinsen L, Bennedsen M, Haaber A, Langholz E, Vegh Z, Duricova D, Jess T, Bell S, Burisch J, Munkholm P. eHealth: individualization of mesalazine treatment through a self-managed web-based solution in mild-to-moderate ulcerative colitis. Inflamm Bowel Dis. 2014 Dec;20(12):2276-85. doi: 10.1097/MIB.0000000000000199. PMID 25248002
- [Background] de Jong MJ, van der Meulen-de Jong AE, Romberg-Camps MJ, Becx MC, Maljaars JP, Cilissen M, van Bodegraven AA, Mahmmod N, Markus T, Hameeteman WM, Dijkstra G, Masclee AA, Boonen A, Winkens B, van Tubergen A, Jonkers DM, Pierik MJ. Telemedicine for management of inflammatory bowel disease (myIBDcoach): a pragmatic, multicentre, randomised controlled trial. Lancet. 2017 Sep 2;390(10098):959-968. doi: 10.1016/S0140-6736(17)31327-2. Epub 2017 Jul 14. PMID 28716313
- [Background] Silverberg MS, Satsangi J, Ahmad T, Arnott ID, Bernstein CN, Brant SR, Caprilli R, Colombel JF, Gasche C, Geboes K, Jewell DP, Karban A, Loftus EV Jr, Pena AS, Riddell RH, Sachar DB, Schreiber S, Steinhart AH, Targan SR, Vermeire S, Warren BF. Toward an integrated clinical, molecular and serological classification of inflammatory bowel disease: report of a Working Party of the 2005 Montreal World Congress of Gastroenterology. Can J Gastroenterol. 2005 Sep;19 Suppl A:5A-36A. doi: 10.1155/2005/269076. PMID 16151544
- [Background] Satsangi J, Silverberg MS, Vermeire S, Colombel JF. The Montreal classification of inflammatory bowel disease: controversies, consensus, and implications. Gut. 2006 Jun;55(6):749-53. doi: 10.1136/gut.2005.082909. PMID 16698746
- [Background] Dignass A, Eliakim R, Magro F, Maaser C, Chowers Y, Geboes K, Mantzaris G, Reinisch W, Colombel JF, Vermeire S, Travis S, Lindsay JO, Van Assche G. Second European evidence-based consensus on the diagnosis and management of ulcerative colitis part 1: definitions and diagnosis. J Crohns Colitis. 2012 Dec;6(10):965-90. doi: 10.1016/j.crohns.2012.09.003. Epub 2012 Oct 3. No abstract available. PMID 23040452
- [Background] Lane ER, Zisman TL, Suskind DL. The microbiota in inflammatory bowel disease: current and therapeutic insights. J Inflamm Res. 2017 Jun 10;10:63-73. doi: 10.2147/JIR.S116088. eCollection 2017. PMID 28652796
- [Background] Hansen JJ, Sartor RB. Therapeutic Manipulation of the Microbiome in IBD: Current Results and Future Approaches. Curr Treat Options Gastroenterol. 2015 Mar;13(1):105-20. doi: 10.1007/s11938-014-0042-7. PMID 25595930
- [Background] Bernstein CN, Forbes JD. Gut Microbiome in Inflammatory Bowel Disease and Other Chronic Immune-Mediated Inflammatory Diseases. Inflamm Intest Dis. 2017 Nov;2(2):116-123. doi: 10.1159/000481401. Epub 2017 Oct 20. PMID 30018962
- [Background] Franzosa EA, Sirota-Madi A, Avila-Pacheco J, Fornelos N, Haiser HJ, Reinker S, Vatanen T, Hall AB, Mallick H, McIver LJ, Sauk JS, Wilson RG, Stevens BW, Scott JM, Pierce K, Deik AA, Bullock K, Imhann F, Porter JA, Zhernakova A, Fu J, Weersma RK, Wijmenga C, Clish CB, Vlamakis H, Huttenhower C, Xavier RJ. Gut microbiome structure and metabolic activity in inflammatory bowel disease. Nat Microbiol. 2019 Feb;4(2):293-305. doi: 10.1038/s41564-018-0306-4. Epub 2018 Dec 10. PMID 30531976
- [Background] Burisch J, Jess T, Martinato M, Lakatos PL; ECCO -EpiCom. The burden of inflammatory bowel disease in Europe. J Crohns Colitis. 2013 May;7(4):322-37. doi: 10.1016/j.crohns.2013.01.010. Epub 2013 Feb 8. PMID 23395397
- [Background] Burisch J, Katsanos KH, Christodoulou DK, Barros L, Magro F, Pedersen N, Kjeldsen J, Vegh Z, Lakatos PL, Eriksson C, Halfvarson J, Fumery M, Gower-Rousseau C, Brinar M, Cukovic-Cavka S, Nikulina I, Belousova E, Myers S, Sebastian S, Kiudelis G, Kupcinskas L, Schwartz D, Odes S, Kaimakliotis IP, Valpiani D, D'Inca R, Salupere R, Chetcuti Zammit S, Ellul P, Duricova D, Bortlik M, Goldis A, Kievit HAL, Toca A, Turcan S, Midjord J, Nielsen KR, Andersen KW, Andersen V, Misra R, Arebi N, Oksanen P, Collin P, de Castro L, Hernandez V, Langholz E, Munkholm P; Epi-IBD Group. Natural Disease Course of Ulcerative Colitis During the First Five Years of Follow-up in a European Population-based Inception Cohort-An Epi-IBD Study. J Crohns Colitis. 2019 Feb 1;13(2):198-208. doi: 10.1093/ecco-jcc/jjy154. PMID 30289522
- [Background] Burisch J, Zammit SC, Ellul P, Turcan S, Duricova D, Bortlik M, Andersen KW, Andersen V, Kaimakliotis IP, Fumery M, Gower-Rousseau C, Girardin G, Valpiani D, Goldis A, Brinar M, Cukovic-Cavka S, Oksanen P, Collin P, Barros L, Magro F, Misra R, Arebi N, Eriksson C, Halfvarson J, Kievit HAL, Pedersen N, Kjeldsen J, Myers S, Sebastian S, Katsanos KH, Christodoulou DK, Midjord J, Nielsen KR, Kiudelis G, Kupcinskas L, Nikulina I, Belousova E, Schwartz D, Odes S, Salupere R, Carmona A, Pineda JR, Vegh Z, Lakatos PL, Langholz E, Munkholm P; Epi-IBD group. Disease course of inflammatory bowel disease unclassified in a European population-based inception cohort: An Epi-IBD study. J Gastroenterol Hepatol. 2019 Jun;34(6):996-1003. doi: 10.1111/jgh.14563. Epub 2019 Jan 21. PMID 30562421
- [Background] Harbord M, Eliakim R, Bettenworth D, Karmiris K, Katsanos K, Kopylov U, Kucharzik T, Molnar T, Raine T, Sebastian S, de Sousa HT, Dignass A, Carbonnel F; European Crohn's and Colitis Organisation [ECCO]. Third European Evidence-based Consensus on Diagnosis and Management of Ulcerative Colitis. Part 2: Current Management. J Crohns Colitis. 2017 Jul 1;11(7):769-784. doi: 10.1093/ecco-jcc/jjx009. No abstract available. PMID 28513805
- [Background] Jarnerot G, Hertervig E, Friis-Liby I, Blomquist L, Karlen P, Granno C, Vilien M, Strom M, Danielsson A, Verbaan H, Hellstrom PM, Magnuson A, Curman B. Infliximab as rescue therapy in severe to moderately severe ulcerative colitis: a randomized, placebo-controlled study. Gastroenterology. 2005 Jun;128(7):1805-11. doi: 10.1053/j.gastro.2005.03.003. PMID 15940615
- [Background] Marin-Jimenez I, Nos P, Domenech E, Riestra S, Gisbert JP, Calvet X, Cortes X, Iglesias E, Huguet JM, Taxonera C, Fernandez R, Carpio D, Gutierrez A, Guardiola J, Laria LC, Sicilia B, Bujanda L, Cea-Calvo L, Romero C, Rincon O, Julia B, Panes J. Diagnostic Performance of the Simple Clinical Colitis Activity Index Self-Administered Online at Home by Patients With Ulcerative Colitis: CRONICA-UC Study. Am J Gastroenterol. 2016 Feb;111(2):261-8. doi: 10.1038/ajg.2015.403. Epub 2016 Jan 12. PMID 26753886
- [Background] Walmsley RS, Ayres RC, Pounder RE, Allan RN. A simple clinical colitis activity index. Gut. 1998 Jul;43(1):29-32. doi: 10.1136/gut.43.1.29. PMID 9771402
- [Background] Bennebroek Evertsz' F, Nieuwkerk PT, Stokkers PC, Ponsioen CY, Bockting CL, Sanderman R, Sprangers MA. The patient simple clinical colitis activity index (P-SCCAI) can detect ulcerative colitis (UC) disease activity in remission: a comparison of the P-SCCAI with clinician-based SCCAI and biological markers. J Crohns Colitis. 2013 Dec;7(11):890-900. doi: 10.1016/j.crohns.2012.11.007. Epub 2012 Dec 24. PMID 23269224
- [Background] Smith LA, Gaya DR. Utility of faecal calprotectin analysis in adult inflammatory bowel disease. World J Gastroenterol. 2012 Dec 14;18(46):6782-9. doi: 10.3748/wjg.v18.i46.6782. PMID 23239916
- [Background] Costa F, Mumolo MG, Ceccarelli L, Bellini M, Romano MR, Sterpi C, Ricchiuti A, Marchi S, Bottai M. Calprotectin is a stronger predictive marker of relapse in ulcerative colitis than in Crohn's disease. Gut. 2005 Mar;54(3):364-8. doi: 10.1136/gut.2004.043406. PMID 15710984
- [Background] Li J, Zhao X, Li X, Lu M, Zhang H. Systematic Review with Meta-Analysis: Fecal Calprotectin as a Surrogate Marker for Predicting Relapse in Adults with Ulcerative Colitis. Mediators Inflamm. 2019 May 28;2019:2136501. doi: 10.1155/2019/2136501. eCollection 2019. PMID 31275056
- [Background] Ankersen DV, Carlsen K, Marker D, Munkholm P, Burisch J. Using eHealth strategies in delivering dietary and other therapies in patients with irritable bowel syndrome and inflammatory bowel disease. J Gastroenterol Hepatol. 2017 Mar;32 Suppl 1:27-31. doi: 10.1111/jgh.13691. PMID 28244677
- [Background] Irvine EJ, Zhou Q, Thompson AK. The Short Inflammatory Bowel Disease Questionnaire: a quality of life instrument for community physicians managing inflammatory bowel disease. CCRPT Investigators. Canadian Crohn's Relapse Prevention Trial. Am J Gastroenterol. 1996 Aug;91(8):1571-8. PMID 8759664
- [Background] Jowett SL, Seal CJ, Barton JR, Welfare MR. The short inflammatory bowel disease questionnaire is reliable and responsive to clinically important change in ulcerative colitis. Am J Gastroenterol. 2001 Oct;96(10):2921-8. doi: 10.1111/j.1572-0241.2001.04682.x. PMID 11693327
- [Background] Ghosh S, Louis E, Beaugerie L, Bossuyt P, Bouguen G, Bourreille A, Ferrante M, Franchimont D, Frost K, Hebuterne X, Marshall JK, O'Shea C, Rosenfeld G, Williams C, Peyrin-Biroulet L. Development of the IBD Disk: A Visual Self-administered Tool for Assessing Disability in Inflammatory Bowel Diseases. Inflamm Bowel Dis. 2017 Mar;23(3):333-340. doi: 10.1097/MIB.0000000000001033. PMID 28146002